CLINICAL TRIAL: NCT06346015
Title: Efficacy of Gamma Entrainment Stimulation for Cognitive Dysfunction After Aneurysmal Subarachnoid Hemorrhage: a Prospective Randomized Controlled Trial
Brief Title: Gamma Entrainment Stimulation for Cognitive Dysfunction After aSAH
Acronym: GES-aSAH
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Collaborators: Shanghai Joyingmed Sensory Stimulation Lab (Unknown)
Responsible Party: Principal Investigator, Xiaolin Chen, MD, Director, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HX-A-2023050
Record Dates: First submitted 2023-12-18; First posted 2024-04-03 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-03

CONDITIONS: Subarachnoid Hemorrhage, Aneurysmal; Cognitive Dysfunction
MeSH Terms: conditions — Subarachnoid Hemorrhage; Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The relevant neuroimaging evaluation process is blinded to the evaluator to ensure the objectivity of the evaluation results.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gamma Entrainment Stimulation + Standard Care (Experimental): Gamma Entrainment Stimulation
  Interventions: Procedure: Gamma Entrainment Stimulation
- Standard Care (No Intervention)

INTERVENTIONS:
Procedure: Gamma Entrainment Stimulation — Audio-assisted therapy: receive audio therapy with a specific device for 30 minutes, once in the morning and evening for 3 months.
  (Binaural beat treatment group: receive binaural beat treatment with a specific device for 30 minutes, once in the morning and evening, for 3 months.）
  Other Names: Audio-assistied therapy
  Arms: Gamma Entrainment Stimulation + Standard Care

SUMMARY:
The goal of this clinical trial is to Explore and verify whether 40Hz audio and binaural beat 40Hz audio can improve the postoperative cognitive dysfunction seen in patients with aneurysmal subarachnoid hemorrhage. This study is a single-center, prospective, randomized, controlled clinical trial. Patients with aneurysmal subarachnoid hemorrhage were selected and randomized into intervention group (audio adjuvant group) and control group (conventional treatment group). Patients in the intervention group will receive audio therapy after surgery, and patients in the control group will receive usual care. EEG, fMRI and mRS scores were evaluated after 3 months of follow-up.

DETAILED DESCRIPTION:
Aneurysmal subarachnoid hemorrhage (aSAH) is a neurological malady that has garnered global public health apprehension due to its severity. Research indicates that cerebral ischemic events subsequent to aSAH treatment are both pervasive and intricate, with their occurrence mechanism and timing categorized into early and late onset. Early cerebral ischemia typically manifests within 1-3 days post-aSAH onset, primarily attributed to factors such as cerebral vasospasm, hemorrhagic cerebral edema, and thrombosis. The severity of these lesions can be alleviated through medical, endovascular, and surgical interventions. Conversely, delayed cerebral ischemia generally arises between 4 days to 2 weeks after surgery, predominantly stemming from cerebral edema, inflammatory reactions, cortical depolarization, and microthrombosis. Managing delayed cerebral ischemia necessitates vigilant patient monitoring and the maintenance of stable cerebral blood flow, achieved by mitigating the impact of cerebral edema and inflammatory responses. Cerebral ischemia induces physiological changes like nerve cell damage, apoptosis, glial cell proliferation, and inflammatory responses, potentially impacting brain function, particularly cognitive function. Consequently, the application of our established TAPS prognostic model effectively identifies individuals at a higher risk of cognitive dysfunction and poor prognosis, facilitating the screening of potential intervention candidates for this study.

In recent years, the scientific community has discerned the pivotal role of microglia in preserving the stability of the brain environment. By modulating their activities, the degree of ischemia can be effectively controlled, mitigating subsequent impairments in brain function. This revelation forms the basis for pioneering nonpharmacological treatment strategies. Among these innovative approaches, frequency-specific audio therapy, notably utilizing 40Hz audio and binaural beat audio, has garnered significant attention. 40Hz audio induces gamma waves in the brain, linked to cognitive functions such as attention, memory, and perception. Binaural beat audio, a neuroacoustic phenomenon, involves introducing two sounds with slightly different frequencies to the ears, prompting the brain to create a new EEG frequency. Regarding 40Hz audio, its potential efficacy is closely tied to the induction of gamma waves, associated with heightened focus and information processing. Laboratory studies suggest that playing 40Hz audio stimulates the brain to produce more gamma waves, hinting at its potential to enhance human cognitive function by regulating electrical brain activity. Binaural beat audio operates on a more intricate level. The brain attempts to "synchronize" two audio pieces with slightly different frequencies, generating a new EEG frequency. This neuroacoustic phenomenon induces specific brain activity, potentially enhancing cognitive function. Crucially, whether 40Hz audio or binaural beat audio, their efficacy may hinge on the "neuroplasticity" of the brain, signifying the brain's ability to alter its structure and function in response to sustained external stimulation. This "frequency-following response" induced by audio stimuli may bring about neuroplasticity changes, further enhancing cognitive function.

For specific brain disorders like Alzheimer's disease, audio therapy could prove impactful. In Alzheimer's patients, gamma-wave activity in the brain is typically diminished, but preliminary studies indicate that 40Hz audio stimulation may enhance gamma activity, potentially improving memory and attention. Moreover, binaural beat audio may contribute to enhancing mental and physical well-being. Research suggests that it can modify the brain's electrical activity pattern, improving emotional states, reducing anxiety and stress, and enhancing sleep quality.

In conclusion, both 40Hz audio and binaural beat audio, as potential non-pharmacological therapeutic strategies, warrant widespread attention from the research community. Although the current study is in its early stages, if audio therapy effectively ameliorates the cognitive dysfunction resulting from aneurysmal subarachnoid hemorrhage, it could introduce novel possibilities for the rehabilitation of this condition.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of aneurysmal subarachnoid hemorrhage and aneurysm secured
2. Postoperative TAPS score ≥ 2 points
3. Age: 18 years old and 75 years old
4. Hearing function is not impaired and audio therapy is well tolerated
5. informed Consented

Exclusion Criteria:

1. Hearing impairment or significant discomfort with audio therapy
2. In other clinical trials within three months before the trial
3. Pregnant women and lactating women
4. Drugs that may affect cognitive function should be used during the study
5. Previous history including cognitive dysfunction or mental illness

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Montreal Cognitive Assessment (MoCA) scores < 22 | at 3 months after enrollment
mini-mental state examiniation (MMSE) < 27 | at 3 months after enrollment
modified Rankin Scales (mRS) > 2 | at 3 months after enrollment
  unfavorable outcome

SECONDARY OUTCOMES:
electroencephalogram (EEG) indicators | at 3 months after enrollment
  auditory steady state evoked response (ASSR) P(50), N(100) and P(200) components Frequency following responses (FFRs) EEG frequency ranges of alpha, beta, delta, theta and gamma
functional Magnetic Resonance Imaging (fMRI) indicators | at 3 months after enrollment
  ALFF: Amplitude of Low Frequency Fluctuation fALFF: fractional Amplitude of Low Frequency Fluctuation ReHo: Regional Homogeneity FC: Functional Connectivity VMHC: Voxel-Mirrored Homotopic Connectivity FCD: Functional Connectivity Density

OTHER OUTCOMES:
Safety indicator | at 3 months after enrollment
  the occurrence of serious adverse events. Including, but not limited to, serious physical or psychological reactions, serious complications or other health problems. All adverse events and serious adverse events will be recorded in detail, including the nature of the event, time to start and end, severity, association with study treatment, management measures, and outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Guangzhi Shi, MD, Study Director — Beijing Tiantan Hospital; Jun Yang, MD, Study Director — Beijing Tiantan Hospital; Yu Chen, MD, Study Director — Beijing Tiantan Hospital; Ke Wang, MD, Study Director — Beijing Tiantan Hospital; Cunyang Li, MD, Study Director — Beijing Tiantan Hospital; Junwei Lv, MD, Study Director — Shanghai Joyingmed Sensory Stimulation Lab; Nianze Chen, MD, Study Director — Shanghai Joyingmed Sensory Stimulation Lab

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Iaccarino HF, Singer AC, Martorell AJ, Rudenko A, Gao F, Gillingham TZ, Mathys H, Seo J, Kritskiy O, Abdurrob F, Adaikkan C, Canter RG, Rueda R, Brown EN, Boyden ES, Tsai LH. Gamma frequency entrainment attenuates amyloid load and modifies microglia. Nature. 2016 Dec 7;540(7632):230-235. doi: 10.1038/nature20587. PMID 27929004
- [Background] Martorell AJ, Paulson AL, Suk HJ, Abdurrob F, Drummond GT, Guan W, Young JZ, Kim DN, Kritskiy O, Barker SJ, Mangena V, Prince SM, Brown EN, Chung K, Boyden ES, Singer AC, Tsai LH. Multi-sensory Gamma Stimulation Ameliorates Alzheimer's-Associated Pathology and Improves Cognition. Cell. 2019 Apr 4;177(2):256-271.e22. doi: 10.1016/j.cell.2019.02.014. Epub 2019 Mar 14. PMID 30879788
- [Background] Adaikkan C, Middleton SJ, Marco A, Pao PC, Mathys H, Kim DN, Gao F, Young JZ, Suk HJ, Boyden ES, McHugh TJ, Tsai LH. Gamma Entrainment Binds Higher-Order Brain Regions and Offers Neuroprotection. Neuron. 2019 Jun 5;102(5):929-943.e8. doi: 10.1016/j.neuron.2019.04.011. Epub 2019 May 7. PMID 31076275
- [Background] Chen X, Shi X, Wu Y, Zhou Z, Chen S, Han Y, Shan C. Gamma oscillations and application of 40-Hz audiovisual stimulation to improve brain function. Brain Behav. 2022 Dec;12(12):e2811. doi: 10.1002/brb3.2811. Epub 2022 Nov 14. PMID 36374520